CLINICAL TRIAL: NCT00153478
Title: Project CHOICES Efficacy Study for Preventing Alcohol-Exposed Pregnancies
Brief Title: Project CHOICES Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-3271
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Risk for an Alcohol-Exposed Pregnancy; Hazardous Alcohol Use; Risk for Unintended Pregnancy
Keywords: Alcohol-Exposed Pregnancy; Binge drinking; Frequent drinking; Unintended pregnancy; Fetal Alcohol Syndrome
MeSH Terms: conditions — Binge Drinking; Fetal Alcohol Spectrum Disorders

INTERVENTIONS:
Behavioral: Brief Motivational Counseling

SUMMARY:
Project CHOICES Efficacy Study is a randomized controlled trial (RCT) designed to evaluate the clinical efficacy of a brief motivational intervention aimed at reducing alcohol-exposed pregnancies(AEP)in high-risk preconceptional women. The study is a multi-site collaborative study between the CDC and three universities. The hypothesis of the study is that a greater proportion of women will reduce thier risk of having an alcohol-exposed pregnancy after participating in the Information Plus Counseling (IPC) intervention than do those in the Information Only(IO) control group.

DETAILED DESCRIPTION:
Women at high risk for an AEP are define as sexually active, fertile women who are drinking more than 7 drinks per week and/or 5 or more drinks on any one day, and are noy using effective measures to prevent pregnancy. Participants will be recruited from community-based setting previously shown to have increased proportions of women at risk for AEP. Women in the intervention group (IPC) will receive 4 counselling sessions that include personal feedback on AEP risk behaviors drawn from baseline information,consequences of alcohol use in pregnancy, assessing readiness to change risk behaviors, pros and cons of risk drinking and unprotected intercourse, goal setting to reduce risk behaviors, and a consultation visit with a family planning provider to discuss appropriate choices for pregnancy prevention based on clinical assessment. Clients are counseled that there are two routes to reducing AEP risk, alcohol reduction or pregnancy prevention, with the ideal being both. Women in the control group (IO) will receive an informational brochure that addresses healthy lifestyle behaviors, including alcohol use, and a list of referral sources for health care treatment and alcohol abuse treatment. Both groups will be assessed at baseline using a full battery of measures that include alcohol and contraceptive use with follow-up measures at 3, 6, and 9 months after baseline.

ELIGIBILITY:
Inclusion Criteria: Women who: are not pregnant, are between the ages of 18 and 44 years, consume more than seven drinks per week and/or at least one binge episode (five or more drinks in one day) in the last 90 days (for the Texas jail & recovery center sites, this will be the 90 days before entering these facilities), are able to provide and do provide informed consent, are members of the special setting's population, and are available for follow-up through 9 months after recruitment.

-

Exclusion Criteria: Women who: do not meet the inclusion criteria, cannot commit to provide information about how to be contacted for follow-up, or are unable to understand spoken English.

-

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200
Dates: Start 2002-07; Study Completion 2004-08

PRIMARY OUTCOMES:
Reduced risks for AEP;reduced risk drinking and reduced episodes of unprotected intercourse.

SECONDARY OUTCOMES:
Mediators and moderators of reduced risk in the IPC and IO groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa L Floyd, DSN, Principal Investigator — Centers for Disease Control and Prevention; Mark B Sobell, PhD, Principal Investigator — Nova Southeastern University; Mary V. Velasquez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Karen Ingersol, PhD, Principal Investigator — Virginia Commonwealth University
Locations (11):
- United States (11):
  - Broward County Health District Primary Care Centers, Fort Lauderdale, Florida
  - Media Recruited Participants from Broward County, Fort Lauderdale, Florida
  - Plane State Jail, Dayton, Texas
  - Career and Recovery, Houston, Texas
  - Door to Recovery, Houston, Texas
  - Harris County Jail, Houston, Texas
  - Houston Recovery Campus, Houston, Texas
  - New Directions, Houston, Texas
  - Sally's House, Houston, Texas
  - Medicaid Helath Maintenance Organization, Richmond, Virginia
  - Outpatient Gynecology Clinic-Virginia Commonwealth Univ, Richmond, Virginia